CLINICAL TRIAL: NCT00849537
Title: The Effect of Intravitral Injection of Triamcinolone Combined With Cataract Surgery (Phacoemulsification) on Diabetic Macular Edema and Diabetic Retinopathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Shaheed Beheshti Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8711
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Diabetic Retinopathy
Keywords: Triamcinolon; Cataract; Diabetic retinopathy; non-proliferative retinopathy
MeSH Terms: conditions — Diabetic Retinopathy; Cataract | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Triamcinolone (Experimental): Injection of intravitreal Triamcinolone
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Triamcinolone — Injection of intravitreal Triamcinolone

SUMMARY:
In this study, regressed proliferative diabetic retinopathy, very severe, severe and moderate non-prolifrative diabetic retinopathy patients who were going to have a cataract surgery, underwent a complete eye examination, OCT, FAG and color photography 2 weeks prior to their operation. All patients divided in two: 1) control group (Phyco,PCIOL), 2) triamcinolone treatment group (Phaco with PCIOL+IVT). One month after surgery a complete eye examination will be done especially; IOP and endophthalmitis. A 6 month follow-up will be done for these two groups and diabetic retinopathy progression will be checked.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with non-proliferative diabetic retinopathy and regressed PDR

Exclusion Criteria:

* Uncontrolled HTN
* History of glaucoma
* Active PDR
* NVI
* TRD
* Any ophthalmic operation
* Renal problem(cr>3)
* CVA
* Uveitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2008-04; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Macula diameter | 6th week, 3, 6 months

SECONDARY OUTCOMES:
Diabetic retinopathy | 6th weeks, 3 and 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Siamak Moradian, MD, Principal Investigator — Shaheed Beheshti University Of Medical Science
Locations (3):
- Iran (3):
  - Ophthalmic Research Centre, Tehran, Tehran Province
  - Siamak Moradian,MD, Tehran, Tehran Province
  - Tehran